CLINICAL TRIAL: NCT04273074
Title: Point of Care Upper Airway Ultrasound in the Assessment of Difficult Visualization of the Larynx in Obese Patients Undergoing Bariatric Surgery: a Comparison With the Conventional Cormack-Lehane Classification During Direct Laryngoscopy: an Observational Study
Brief Title: Upper Airway Ultrasound in the Assessment of Difficult Visualization of the Larynx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D-18-2019
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Airway Assessment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- preoperative sonographic assessment group (Other): preoperative sonographic assessment to airway
  Interventions: Radiation: sonographic assessment

INTERVENTIONS:
Radiation: sonographic assessment — preoperative sonographic assessment to airway

SUMMARY:
failed and Difficult tracheal intubation after direct laryngoscopy is a dreaded complication of general anesthesia as it is associated with serious morbidity and mortality. There are several conventional clinical airway assessment parameters such as the modified Mallampati classification,thyromental and hyomental distance, interincisor distance, neck movementsand neck circumference, which are usually used to predict a difficult airwayand are components of multivariate risk indices. Despite the use of these parameters, the diagnostic accuracy of a preanesthetic airway assessment in predicting difficult intubation is very low. Ultrasound has been evolving as a useful device for airway assessment,and sublingual ultrasound has been used for this purpose.

DETAILED DESCRIPTION:
By an anesthesiologist who is experienced in airway ultrasound, patients will preoperative sonographic assessment . the patient will lie in the ramped up position , with head in the neutral position.The linear probe of the ultrasound machine will be used. Under the patient's chin, The probe of ultrasond will be placed , at different levels, to get the of the submandibular area in transverse view and the upper part of the neck. The transverse view will be used for measuring the the skin to hyoid, tongue volume,and the skin to epiglottis distance. The mid-sagittal view will be used for measuring the distance between epiglottis ,pre-epiglottic space , vocal cords, and the neck fat volume .

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients above 18 years of age.
2. Both genders
3. Patients scheduled for elective surgery under general anesthesia
4. Obese patients with BMI > 30 kg/m2

Exclusion Criteria:

1. Patients with psychological disorders or those lacking co-operation.
2. Patients with maxillofacial anomalies, restricted neck movements and limited mouth opening.
3. American Society of Anesthesiologists (ASA) physical status class IV
4. Emergency operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Epiglottis-to-vocal-cord distance | during examination up to 1 hours
  Epiglottis-to-vocal-cord distance by ultrasound

SECONDARY OUTCOMES:
Tongue width | UP TO 1 HOURE
  by ultrasound
Modified Mallampati class | UP TO 1 HOURE
  Class I: Soft palate, fauces, pillars, and uvula are visible.
  Class II: Soft palate, fauces, and uvula are visible.
  Class III: Soft palate and base of uvula are visible.
  Class IV: Soft palate is not visible at all.
  Class I and II were defined as "good view" and III and IV as "poor view" in the present study.
the time needed to perform the ultrasound examination. | UP TO 1 HOURE
  by minute
Pre-epiglottic space | UP TO 1 HOURE
  by ultrasound
Pre-epiglottic space | up to 1 hour
  by ultrasound
Skin to hyoid distance | up to 1 hour
  by ultrasound
Skin to epiglottis distance | up to 1 hour
  by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Helmy, MD, Principal Investigator — Professor of Anaesthesia, surgical ICU &Pain management; Yasmine salah, Principal Investigator — lecturer of Anesthesiology
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still working